CLINICAL TRIAL: NCT01587508
Title: A Phase III, Randomized, Single-Blind, Superiority Study Comparing The Efficacy And Tolerability Of A New Drug Containing The Combination Meloxicam And Cyclobenzaprine And The Same Components Alone In The Treatment Of Acute Lumbago
Brief Title: Study Comparing A New Drug Containing The Combination Meloxicam And Cyclobenzaprine In The Treatment Of Acute Lumbago
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The comparator product was withdrawn from the brazilian market not being possible to conduct the design regarding initially planned.
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EF 127
Record Dates: First submitted 2012-04-24; First posted 2012-04-30 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2012-04

CONDITIONS: Acute Lumbago
MeSH Terms: interventions — Meloxicam; cyclobenzaprine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- meloxicam - Movatec® (Active Comparator)
  Interventions: Drug: meloxicam - Movatec®
- cyclobenzaprine - Miosan®, (Active Comparator)
  Interventions: Drug: cyclobenzaprine - Miosan®
- meloxicam/cyclobenzaprine hydrochloride (Experimental)
  Interventions: Drug: meloxicam/cyclobenzaprine hydrochloride

INTERVENTIONS:
Drug: meloxicam/cyclobenzaprine hydrochloride — two oral capsules a day during approximately 07 days
  Arms: meloxicam/cyclobenzaprine hydrochloride
Drug: meloxicam - Movatec® — two oral tablet a day during approximately 07 days
  Arms: meloxicam - Movatec®
Drug: cyclobenzaprine - Miosan® — two oral tablet a day during approximately 07 days
  Arms: cyclobenzaprine - Miosan®,

SUMMARY:
The purpose of this study is to assess the efficacy end tolerability of a new drug containing the combination meloxicam and cyclobenzaprine (7,5/10mg) and the same components alone in the treatment of acute lumbago.

DETAILED DESCRIPTION:
To assess the efficacy and tolerability of a new drug containing the combination meloxicam and cyclobenzaprine in the treatment of acute lumbago, compared to the same components alone.

Some eligibility criteria:

Have a normal X-ray of the lumbar spine for the age; Have a baseline score in the VAS higher than or equal to 40 mm

ELIGIBILITY:
Inclusion Criteria:

* Sign, initial and date the Informed Consent Form (ICF);
* Be between 18 and 75 years old;
* Have acute lumbago with onset in less than 72 hours;
* Have a normal X-ray;
* Have a baseline score in the VAS higher than or equal to 40 mm;

Exclusion Criteria:

* Use of triptans;
* Use of monoamine oxidase inhibitors;
* Use of NSAIDs within the last week;
* Previous use of narcotics;
* Have any rheumatologic disease;
* Conditions of chronic pain;
* Have any significant chronic comorbidity;
* Previous history of gastrointestinal bleed or ulcers;
* History of allergy to any of the components of study medications;
* Recent history of a myocardial infarction, cardiac arrhythmia, cardiac conduction block or change, or congestive heart failure;
* Female patients who are pregnant or breastfeeding or who wish to become pregnant or who deny using safe contraceptive methods during the study will not be enrolled in the study;
* Have participated in another clinical trial within the last 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | Pain reduction 3 days after the administration of study drugs
  Compare the treatment groups for the efficacy in pain reduction, 3 days after the administration of study drugs, when compared to the baseline assessment.

SECONDARY OUTCOMES:
Frequency of rescue medication use | During study treatment, an expected average of 7days
  Assessment of frequency of rescue medication use, as well as the proportion of patients during study treatment;

CONTACTS AND LOCATIONS:
Overall Officials: Alceu Chueiri, Principal Investigator — Hospital de Base de São José do Rio Preto; Paulo Guilherme, Principal Investigator — Hospital Santa Marcelina; Wagner Caiafa, Principal Investigator — Santa Casa de Juiz de Fora; Antonio Scotton, Principal Investigator — Centro MIneiro de Pesquisa - Juiz de Fora; Lindomar G. Oliveira, Principal Investigator — Clínica de Ortopedia e Fraturas de Goiania; Antonio Carlos Ximenes, Principal Investigator — CIP Pesquisas Médicas Ltda; Sonia Alvarenga, Principal Investigator — Faculdade de Medicina ABC; Gilberto Brandão, Principal Investigator — Clínica Perdizes; Luciana Teixeira, Principal Investigator — IMA Brasil - Instituto de Medicina Avançada; Antonio Tarcísio, Principal Investigator — Santa Casa de Misericórdia de Belo Horizonte; Carlos Roberto Galia, Principal Investigator — Hospital de Clínicas de Porto Alegre; Mauro Hernandes, Principal Investigator — Santa Casa de Votuporanga
Locations (11):
- Brazil (11):
  - CIP Pesquisas Médicas Ltda, Goiânia, Goiás
  - Clínica de Ortopedia e Fraturas de Goiânia, Goiânia, Goiás
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Santa Casa de Juíz de Fora, Juiz de Fora, Minas Gerais
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina ABC, Santo André, São Paulo
  - Hospítal de Base, São José Rio Preto, São Paulo
  - Clinica de Ortopedia e Fisiatria Perdizes, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - IMA Brasil, São Paulo, São Paulo
  - Santa Casa de Votuporanga, Votuporanga, São Paulo